CLINICAL TRIAL: NCT06325319
Title: Effectiveness of Community Engagement Using M-Mama Champions in Improving Literacy of Obstetric Danger Signs, Birth Preparedness and Complication Readiness Among Pregnant Women in Bahi, Dodoma
Brief Title: Effect of Community Engagement Using M-Mama Champions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dodoma (Other)
Collaborators: Stephen Kibusi (Unknown); James Tumaini Kengia (Unknown)
Responsible Party: Principal Investigator, Alex Sanga, Doctor, University of Dodoma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Ref. No. MA.84/261/02/1/115
Record Dates: First submitted 2024-03-06; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Obstetric Complication; Woman's Role
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-MAMA Champions group (Experimental): Those study participants randomized to the intervention arm will receive the intervention being tested in this study. The intervention will be community engagement through the M-MAMA Champions on obstetric danger signs, birth preparedness, and complication readiness, whereby sensitization to pregnant women will be done. The sensitization package will be delivered by M-MAMA Champions and will encompass obstetric danger signs, birth preparedness, and complication readiness that will be adapted from the Ministry of Health, Tanzania. The package is being used to empower Community Health Workers (CHWs). The intervention is expected to be delivered in two (2) wards (4 Clusters) to be selected in Bahi Council, Dodoma for a period of one month from March to April 2024 and raise awareness by at least 20% in the intervention arm within a study period.
  Interventions: Other: Community engagement using M-MAMA Champions to improve awareness on obstetric danger signs, bith preparedness and complication readiness among pregnant women
- Routine service group (No Intervention): The study participants who will be randomized to the control arm won't receive the intervention, instead, they will continue receiving the routine services. The routine services for pregnant women specifically on knowledge-related empowerment include the package delivered by the healthcare workers at the reproductive and child health clinics. The package is delivered during every Ante Natal Care (ANC) visit to the pregnant woman. The package contains basic information that is also tailored to the specific needs of pregnant women and is delivered with much emphasis to those who are prone to experience pregnancy-related complications for instance, those with Bad Obstetric History (BOH), cardiovascular diseases, or diabetics. The control groups are expected to be derived from two (2) wards (4 Clusters) to be selected in Bahi Council, Dodoma

INTERVENTIONS:
Other: Community engagement using M-MAMA Champions to improve awareness on obstetric danger signs, bith preparedness and complication readiness among pregnant women — Community engagement using M-MAMA Champions to improve awareness of obstetric danger signs, birth preparedness, and complication readiness among pregnant women. The empowered M-MAMA Champions will deliver the intervention to pregnant women in their communities. A total of three (3) sessions will be held, whereby each will take two (2) hours. The sensitization will take place at one of the study participant's residential area, where women will gather up and be sensitized on the subject by the M-MAMA Champion as a facilitator using a well-prepared brochure (package).
  Other Names: Educational intervention
  Arms: M-MAMA Champions group

SUMMARY:
This study aims to determine the effectiveness of community engagement using M-MAMA Champions on awareness of Obstetric Danger Signs, Birth Preparedness, and Complication Readiness among Pregnant Women in Bahi, Dodoma. This is a community-based, cluster randomized controlled trial (cRCT) study, whereby 120 first and second-trimester pregnant women will be randomized at a ratio of 1:1 to the intervention and control groups. The intervention of sensitizing pregnant women on Obstetric danger signs, birth preparedness, and complication readiness by the empowered M-MAMA Champions to the intervention arm clusters will be done for one month, a two-hour session will be delivered every two weeks, using participatory learning and action model for women groups to test the effectiveness of M-MAMA Champions in improving literacy level of obstetric danger signs, birth preparedness and complication readiness and its practice among pregnant women.

The following is the hypothesis being tested

Null Hypothesis; There is no difference in improvement of awareness of Obstetric Danger Signs, Birth Preparedness, and Complication Readiness among Pregnant Women when community engagement is done using M-MAMA Champions compared to routine approaches.

Alternative hypothesis; Community engagement using M-MAMA Champions to improve awareness of Obstetric Danger Signs, Birth Preparedness, and Complication Readiness among Pregnant Women is more effective than routine approaches.

During each 2-hour session, five (5) women will gather up and discuss the obstetric danger signs, birth preparedness, and complication readiness with the assistance of the M-MAMA Champion as a facilitator. An approved brochure on the concerned subject will be used for sensitization. Baseline data will be collected before and after the intervention.

The control arm won't receive any intervention.

DETAILED DESCRIPTION:
Introduction:

Maternal mortality remains a global public health issue, Sustainable Development Goal (SDG) 3 targets to reduce it to less than 70 for every 100,000 live births by 2030 globally. Maternal mortality whose peak is during intrapartum and the first day post-partum, 75% of it is accounted for by obstetric danger signs complications. Tanzania's maternal mortality ratio stands at 104 for every 100,000 live births, higher than the SDG target. Innovations that include women groups like M-MAMA Champions are necessary to improve the literacy level of obstetric danger signs, birth preparedness, and complication readiness among pregnant women and enhance obstetric emergency response and service utilization, for essential interventions in healthcare facilities alone haven't been able to reduce maternal mortality due to poor services utilization.

Methods and analysis:

A community-based, cluster randomized controlled trial (cRCT) design, will be utilized in undertaking the study of 120 first and second-trimester pregnant women randomized at a ratio of 1:1 to the intervention and control groups. The intervention of sensitizing pregnant women on Obstetric danger signs, birth preparedness, and complication readiness by the empowered M-MAMA Champions to the intervention arm clusters will be done for one month, each two-hour session delivered in two weeks, using participatory learning and action model for women groups. The effect of the intervention will be determined using repeated ANOVA analysis.

Ethics and dissemination. The University of Dodoma Research Ethics Committee approved this study (Ref. No. MA.84/261/02/1/115). The study will ensure the protection of the participants' values, dignity, and integrity by the Helsinki Declaration by the World Medical Association. The study results will be published in peer-reviewed journals and disseminated at various conferences, and the government through the Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the first and second trimester (up to 28 weeks of GA).

Exclusion Criteria:

* Pregnant women who will be sick and admitted,
* Mentally incompetent, and
* Those who won't consent to participate in the study.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in scores from a semi-structured interviewer-administered questionnaire on awareness of obstetric danger signs among pregnant women. | One month (4weeks)
  Change of pregnant women's scores from a semi-structured interviewer-administered questionnaire on the awareness of the obstetric danger signs. It's anticipated that there will be a positive change in scores after the intervention.
Improvement in scores from a semi-structured interviewer-administered questionnaire of awareness of birth preparedness and complication readiness among pregnant women | One month (4weeks)
  Change of pregnant women's scores from a semi-structured interviewer-administered questionnaire on awareness of birth preparedness and complication readiness after the intervention. It's anticipated that the majority will be able to name at least three (3) of five (5) key elements of birth preparedness and complication readiness after the intervention.

SECONDARY OUTCOMES:
Improvement in scores from a semi-structured interviewer-administered questionnaire on reported practice of birth preparedness and complication readiness | One month (4weeks)
  Change in the scores from a semi-structured interviewer-administered questionnaire on the reported practice of birth preparedness and complication readiness among pregnant women after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: James T Kengia, PhD, Study Director — University of Dodoma
Locations (1):
- University of Dodoma, Dodoma, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2moths

REFERENCES:
- [Derived] Sanga A, Kibusi S, Kengia JT. The effectiveness of community engagement using M-Mama champions in improving awareness of obstetric danger signs, birth preparedness and complication readiness among pregnant women in Bahi, Dodoma: A cluster randomized pragmatic implementation trial. PLOS Glob Public Health. 2025 Apr 8;5(4):e0004315. doi: 10.1371/journal.pgph.0004315. eCollection 2025. PMID 40198615